CLINICAL TRIAL: NCT01969383
Title: COMPARATIVE ANALYSIS BETWEEN THE ELECTRICAL ACTIVITY WITH AND WITHOUT MUSCULAR STRENGTH IN WATER AND SOIL
Brief Title: Comparative Analysis Between Electrical Muscle Activity In Water And Soil
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Vale do Paraíba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 06708912.8.0000.5503.
Record Dates: First submitted 2013-10-17; First posted 2013-10-25 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Healthy Individuals.
Keywords: healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- heated pool (Experimental): After selection, all volunteers will be asked to attend two exercise protocols performed on the ground and in the heated pool and the minimum interval of 24 hours between each protocol. Data collection will be performed only with the dominant member of each volunteer.
  Interventions: Other: Heated pool training

INTERVENTIONS:
Other: Heated pool training

SUMMARY:
Muscle activity in the aquatic environment was investigated while performing different exercises by electromyography analysis, due to conflicting results in the literature in relation to the floor. This study evaluated and compared the electrical activity of the rectus femoris and biceps femoris, in aquatic method and on the floor, during flexion and knee extension exercises with and without load.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 35
* Sedentary (who engage in physical activity more than twice a week).

Exclusion Criteria:

* History of pain, trauma and / or surgery on the knee joint;
* Presence of musculo - skeletal

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
COMPARATIVE ANALYSIS BETWEEN THE ELECTRICAL ACTIVITY WITH AND WITHOUT MUSCULAR STRENGTH IN WATER AND SOIL | April-October 2013
  It is believed that there is a decrease in muscle electrical activity following the exercises without resistance in the heated water in comparison with cold water and soil due to muscle relaxation and a reduction of the viscosity of water. Considering the resistance exercises, it is believed that there is an increase in muscle electrical activity when held in cold water in comparison with heated water and soil due to the increased viscosity of water.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda P Silva Lima, Doutora, Principal Investigator — Rehabilitation Engineering Laboratory sensorineural motor
Locations (1):
- Izabela dos Santos Mendes, São José dos Campos, São Paulo, Brazil